CLINICAL TRIAL: NCT03572374
Title: Breast Cancer and the Workforce: Talking to Employers and Medical Staff About Work (TEAMWork)
Brief Title: Talking to Employers and Medical Staff About Breast Cancer Treatment and Your Job
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-217
Record Dates: First submitted 2018-06-08; First posted 2018-06-28 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: Workforce; Employers; Talking to Employers and Medical Staff About Work (TEAMWork); 18-217
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEAMWork App (Experimental): The 2-pronged approach of the intervention is operationalized through 2 menus, 1 focused on interactions with the employer and the other with the clinic team. Each menu has a list of features from which participants can choose to learn about a particular topic. A "My notes" button allows participants to take notes directly on the app. These notes will not be available to the research team, such that participants may use the tool without concerns about privacy. The workplace accommodations menu includes sample videos using trained actors to demonstrate how to approach an employer to request accommodations. Additional features include suggestions for accommodations that may be helpful, templates for letters participants can use when requesting accommodations, links to relevant websites, information about legal protections, and contact information for lawyers and firms that provide pro bono assistance.
  Interventions: Other: TEAMWork App
- Information Booklet (control) (Active Comparator): Participants will receive a booklet that includes the information in the app that can practicably be converted to paper. These participants will not have access to the multimedia aspects of the intervention, such as the videos, but they will have all of the relevant information in the app described above, including suggestions for accommodations, written templates for letters, links to websites, information about legal protections, and contact information for pro bono legal assistance. The booklet will also contain information about chemotherapy, radiation therapy and surgery, recommendations for management of common symptoms, and advice for communicating with the clinic team. The information booklet will be provided entirely on paper, although participants may independently access websites recommended in the booklet. The booklet content will mirror the app with regard to cultural responsiveness and appropriateness for different job types and characteristics.
  Interventions: Other: Information Booklet

INTERVENTIONS:
Other: TEAMWork App — The 2-pronged approach of the intervention is operationalized through 2 menus, 1 focused on interactions with the employer and the other with the clinic team. Each menu has a list of features from which participants can choose to learn about a particular topic. A "My notes" button allows participants to take notes directly on the app. These notes will not be available to the research team, such that participants may use the tool without concerns about privacy. The workplace accommodations menu includes sample videos using trained actors to demonstrate how to approach an employer to request accommodations. Additional features include suggestions for accommodations that may be helpful, templates for letters participants can use when requesting accommodations, links to relevant websites, information about legal protections, and contact information for lawyers and firms that provide pro bono assistance.
  Other Names: Talking to Employers and Medical Staff About Work (TEAMWork)
  Arms: TEAMWork App
Other: Information Booklet — Participants in the control arm will receive a booklet that includes the information in the app that can practicably be converted to paper. These participants will not have access to the multimedia aspects of the intervention, such as the videos, but they will have all of the relevant information in the app described above, including suggestions for accommodations, written templates for letters, links to websites, information about legal protections, and contact information for pro bono legal assistance. The booklet will also contain information about chemotherapy, radiation therapy and surgery, recommendations for management of common symptoms, and advice for communicating with the clinic team. The information booklet will be provided entirely on paper, although participants may independently access websites recommended in the booklet. The booklet content will mirror the app with regard to cultural responsiveness and appropriateness for different job types and characteristics.
  Arms: Information Booklet (control)

SUMMARY:
The purpose of this study is learn more about how being treated for breast cancer affects patients' employment. Researchers are testing an early version of a mobile app designed to help breast cancer patients keep their jobs during and after treatment. The app provides advice for patients to use when having conversations about breast cancer with their employers and their doctors. The app is called TEAMWork (Talking to Employers And Medical staff about Work). In this study, the investigators are asking breast cancer patients who are about to receive treatment or who are currently receiving treatment to tell us what aspects of the app work well, so that they can learn how to improve it.

ELIGIBILITY:
Inclusion Criteria:

Patient Usability Testing Inclusion Criteria:

* History of a cancer diagnosis
* At least 18 years of age
* Male or Female
* The ability to give informed consent in English or Spanish
* Able to use and read a smartphone (iPhone or Android)
* Has a smartphone (iPhone or Android)

Community Usability Testing Inclusion Criteria:

* At least 18 years of age
* Male or Female
* The ability to give informed consent in English or Spanish
* Able to use and read a smartphone (iPhone or Android)
* Has a smartphone (iPhone or Android)

Focus Group and Interview Inclusion Criteria:

* Completed chemotherapy treatment for stage I-III breast cancer.
* Age 18 to 64 (inclusive)
* Female
* Paid employment (full time or part time) in the three months prior to diagnosis or at time of consent to MSK protocol #10-071 (PI: Blinder)
* The ability to give informed consent in English or Spanish
* Able to use and read a smartphone (iPhone or Android)
* Has a smartphone (iPhone or Android)

For Cohort 2:

* Participants was covered by Emergency Medicaid at the time of diagnosis and/or at any point during their treatment for breast cancer

RCT Inclusion Criteria:

* Localized invasive breast cancer (not stage 0 or stage IV) per EMR or breast cancer (not stage 0 or stage IV) per self-report for community participants

  * If electronic medical record does not specify stage and patient is undergoing (neo)adjuvant chemotherapy, assume stage is I, II or III
* Planning to undergo or undergoing adjuvant or neoadjuvant chemotherapy per EMR or planning to undergo or undergo chemotherapy per self-report for community participants
* Age 18 to 64 (inclusive)
* Female
* Employment statue of (full time or part time) (those who are on disability leave/medical leave, and other unique employment circumstances at the PI's dicretion are eligible)
* Language preference as English or Spanish
* Able to use and read a smartphone or tablet (e.g. iPad, iPhone or Android)
* Has access to a smartphone or tablet (e.g. iPad, iPhone or Android)

Exclusion Criteria:

RCT Exclusion Criteria:

* Stage 0 breast cancer (DCIS only)
* Stage IV (metastatic) breast cancer
* Recurrence with metastases of breast cancer
* Participants or family members who are participating in MSK IHCD studies related to social determinants of health

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Enrollment: 546 (Estimated)
Dates: Start 2018-06-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
number of participants still employed | 2 years
  Talking to Employers and Medical Staff About Work (TEAMWork) the mobile application (app) is designed to educate patients and improve their communication skills with their employers and their oncology providers, thereby increasing access to work accommodations and optimizing symptom control during treatment. By increasing patients" ability to work during treatment, we believe the app will help them retain their jobs.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Blinder, M.D., M.Sc., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Memorial Sloan Kettering Basking Ridge (Consent and Follow-up), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent and Follow-up), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and Follow up), Montvale, New Jersey
  - Memorial Sloan Kettering Westchester (Consent and Follow-up), Harrison, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Bellevue Hospital Center (Data Collection Only), New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lincoln Medical and Mental Health Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York

REFERENCES:
- [Derived] Blinder VS, Patil S, Finik J, Makower D, Muppidi M, Lichtenthal WG, Parker PA, Claros M, Suarez J, Narang B, Gany F. An interactive mobile application versus an educational booklet to promote job retention in women undergoing adjuvant chemotherapy for breast cancer: a randomized controlled trial. Trials. 2022 Oct 3;23(1):840. doi: 10.1186/s13063-022-06580-7. PMID 36192754
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm